CLINICAL TRIAL: NCT06270849
Title: Validity and Reliability of the Translated International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms Long Form (ICIQ-FLUTS-LF) in Thai Version and Correlation With the IPSS
Brief Title: Validity and Reliability of ICIQ-FLUTS LF in Thai Version and Correlation With IPSS
Status: Completed | Type: Observational
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Valeerat Swatesutipun, Principle investigator, Thammasat University Hospital
Other Study IDs: MTU-EC-SU-0-002/66
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Validity of Thai Version of the ICIQ-FLUTS LF Questionnaire; Reliability of Thai Version of the ICIQ-FLUTS LF
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female with LUTS: Females who has symptoms of lower urinary tract symptoms
  Interventions: Other: Questionnaire
- Normal control group: Females who no history of LUTS or urinary tract disease
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire to assess severity of LUTS in women.

SUMMARY:
The investigators recruited participants, who were female with LUTS 50 participants for known group validity and 80 normal control females to evaluate for construct validity and test for reliability by statistical analysis.

DETAILED DESCRIPTION:
50 females with LUTS will completed the ICIQ-FLUTS and IPSS and then again at 2 weeks apart to test for convergent validity and test-retest validity.

The normal control group 80 women will completed ICIQ-FLUTS LF for test of construct validity.

ELIGIBILITY:
Inclusion Criteria:

* age at or over 18 years old
* can read and understand Thai language
* have lower urinary tract symptoms

Exclusion Criteria:

* those who have a diagnosis of calculi, urinary tract cancer

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females with lower urinary tract symptoms who can read and understand Thai language.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
How well the ICIQ-FLUTS LF questionnaire in the Thai version can differentiate between females with LUTS and normal females, was assessed by the construction validity. | 10-12 months
  Incontinence Questionnaire - Female Lower Urinary Tract Symptoms Long Form (ICIQ-FLUTS-LF) was divided into 6 subgroups of symptoms measurement, which were storage, voiding, incontinence, bladder pain, post micturition, and ability to stop voiding. The construct validity was determined by comparing the ICIQ-FLUTS LF scores of the target group with the ICIQ-FLUTS LF scores of the control group. The comparisons were performed using the Wilcoxon signed-rank test.
The correlation between items within a subscale of the ICIQ-FLUTS LF questionnaire assessed by internal consistency. | 10-12 months
  The internal consistency (a parameter that verifies correlations between items within a subscale of the questionnaire) was assessed by using Cronbach's alpha coefficients. The assessment was done in each subscale of the questionnaire. If Cronbach's alpha coefficients were between 0.7 and 0.95, the instrument was considered to have good internal consistency.
The consistency of the repeated measurements by the Thai version of the ICIQ-FLUTS LF was assessed by the test-retest reliability. | 10-12 months
  The test-retest reliability (a property of producing repeated measurements that are consistent) was verified by having the participants of the target group answer the questionnaire twice with an interval of 2 weeks between the evaluations. We calculated test-retest reliability by using weighted kappa (κ).

SECONDARY OUTCOMES:
The correlation between the IPSS questionnaire and ICIQ-FLUTS LF questionnaire was assessed by convergent validity. | 10-12 months
  The convergent validity (how closely a test is related to other tests that measure the same or similar constructs) was determined by comparing the ICIQ-FLUTS LF scores of the target group with a known validated questionnaire. In this study we used the International Prostate Symptom Score (IPSS) as the comparison test. The comparisons were performed using Pearson's correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Valeerat Swatesutipun, MD, Principal Investigator — Thammasat University Hospital
Locations (1):
- Thammasat University Hospital, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No